CLINICAL TRIAL: NCT04941300
Title: CRC-HUB-SPOKE: A ColoRectal Cancer Screening Hub for Southern California Community Health Centers
Brief Title: ColoRectal Cancer Screening for Southern California Community Health Centers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Elena Martinez, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: IRB # 190990; 5UH3CA233314-05 (NIH)
Record Dates: First submitted 2021-06-18; First posted 2021-06-28 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Cancer
Keywords: screening; underserved populations
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mailed FIT Outreach (Other): Primer, FIT Kit, Reminders, Abnormal FIT Follow-up
  Interventions: Other: Mailed FIT Outreach; Other: Standardized navigation
- Usual Care (No Intervention)

INTERVENTIONS:
Other: Mailed FIT Outreach — We will mail an introductory letter to eligible individuals describing the importance of CRC screening and noting that follow-up mail will include a FIT Kit. Two weeks later they will receive a packet via mail containing the FIT kit, a one-page invitation inviting FIT completion and FIT instructions, COVID-19 messaging, and a postage-paid envelope for return.
  Arms: Mailed FIT Outreach
Other: Standardized navigation — The standardized navigation includes, but is not limited to, the following key components:
  1. Identification of individuals with abnormal FIT
  2. Results review and colonoscopy order by provider
  3. Results reporting to patient
  4. Insurance approval for colonoscopy
  5. Colonoscopy scheduling
  6. Bowel preparation & colonoscopy completion
  7. Colonoscopy results provided to patient and CHC
  8. Referral-to-Care for patients with CRC (if necessary)
  Arms: Mailed FIT Outreach

SUMMARY:
Colorectal cancer (CRC) screening can reduce cancer deaths. However, screening and abnormal test follow-up rates are low among underserved populations. The screening rates of 19-58%, and rates of colonoscopy completion after abnormal stool tests of 18-57% in community health centers (CHC) systems are low. This highlights an opportunity to improve early detection and decrease burden of CRC in our region. Mailed outreach and navigation programs have been shown to increase colonoscopy completion rate. The next step is to understand how to best implement these programs in the community on a larger scale. To achieve this goal, the investigators propose a Hub-and-Spoke intervention combining centralized strategies to maximize CRC screening, follow-up, and referral-to-care. The investigators hypothesize that this intervention will be superior to usual care for increasing CRC screening, abnormal test follow-up, and referral-to-care.

The investigators will conduct a randomized trial to determine effectiveness in: 1) improvement in proportion of individuals up-to-date with screening 3 years post implementation; 2) proportion with abnormal FIT who complete diagnostic colonoscopy within 6 months; and 3) proportion with CRC completing first treatment evaluation.

The investigators will also evaluate the implementation, scalability, and sustainability of the multi-level implementation strategy. The intervention consists of: Mailed FIT and Reminders. Eligible individuals will receive an introductory letter describing the importance of CRC screening and noting that follow-up mail will include a FIT Kit. It will also be offered to patients who completed prior mailed FIT with normal test results. All materials will be in English and Spanish. Two weeks later, participants will receive a packet via mail containing the FIT kit, a one-page invitation inviting FIT completion and FIT instructions, a postage-paid envelope for return to the patient's CHC, and COVID-19 message. For non-compliant individuals not returning the kit, a reminder phone call and text message will be delivered 2 weeks later. The investigators will track returned letters, individuals who are later found to be up-to date with screening, and those who decline screening. The CHC will provide care coordination for patients with an abnormal FIT result.

ELIGIBILITY:
Mailed FIT Inclusion Criteria:

* Patient had an office visit within the last 12 months at one or more of your health centers. (Use Uniform Data System [UDS] criteria for an office visit.)
* Not up to date with colorectal cancer screening according to the standard UDS query
* Male or Female
* 50 - 75 years old
* Current VALID address in San Diego or Riverside Counties (addresses with a PO box or General Delivery are acceptable)
* Valid Phone Number
* Insured patients only (e.g., Medicare, Medi-Cal, or private insurance)

Exclusion Criteria:

* Absence of a phone number listed in the Electronic Health Record/Electronic Medical Record (EMR)
* Absence of a valid mailing address (e.g. blank field)
* Uninsured
* Patients with a diagnosis or past history of total colectomy or colorectal cancer per UDS criteria.
* Duplicate patients within a health center organization. (If a patient was seen at multiple locations within the past year, only include the patient in the sample for the site where the patient was seen last)

Care Coordination for Abnormal FIT results, add the following to the inclusion criteria:

* Completion of a FIT for Colorectal Cancer Screening during the designated time period
* Abnormal FIT result received and documented in EMR during the designated time period

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55999 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Screening up-to-date (primary) | Three years
  Proportion of age-eligible patients with clinic visit in measurement year up-to-date with screening (FIT or FOBT in prior 12 months, sigmoidoscopy in last 5 years, colonoscopy in last 10 years).
Colonoscopy after abnormal FIT (primary) | Six months
  Proportion of patients with abnormal FIT who complete colonoscopy within 6 months

SECONDARY OUTCOMES:
FIT Completion | Twelve months
  Proportion of patients who have FIT ordered as part of usual care or interventions who complete FIT within 12 months
Time to colonoscopy after abnormal FIT | From date of abnormal FIT results until the date of colonoscopy completion, assessed up to 3 years
  Median time to colonoscopy completion after abnormal FIT
Follow-up process | From date of abnormal FIT results until the date of follow-up process is completed if a CRC is found, assessed up to 3 years
  Proportion of patients with abnormal FIT with a) colonoscopy ordered; b) insurance approval completed; c) precolonoscopy visit scheduled; d) precolonoscopy visit completed; e) adequate bowel preparation at time of colonoscopy; f) treatment evaluation referral initiated and first visit completed if CRC found.

OTHER OUTCOMES:
Repeat screening (exploratory outcome) | 12-14 months
  Proportion of patients who complete one normal FIT with repeat FIT within12-14 months.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Elena Martinez, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, Moores Cancer Center, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Castaneda SF, Gupta S, Nodora JN, Largaespada V, Roesch SC, Rabin BA, Covin J, Ortwine K, Preciado-Hidalgo Y, Howard N, Halpern MT, Martinez ME. Hub-and-Spoke centralized intervention to optimize colorectal cancer screening and follow-up: A pragmatic, cluster-randomized controlled trial protocol. Contemp Clin Trials. 2023 Nov;134:107353. doi: 10.1016/j.cct.2023.107353. Epub 2023 Oct 5. PMID 37802222